CLINICAL TRIAL: NCT00070993
Title: Clinical Trial of Creatine in Amyotrophic Lateral Sclerosis
Brief Title: Creatine for the Treatment of Amyotrophic Lateral Sclerosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Collaborators: Office of Dietary Supplements (ODS) (NIH)
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: R01AT000967-01 (NIH)
Record Dates: First submitted 2003-10-09; First posted 2003-10-13 (Estimated); Last update posted 2006-08-04 (Estimated); Status verified 2006-08

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: ALS; Creatine
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — Creatine

INTERVENTIONS:
Drug: creatine monohydrate

SUMMARY:
Creatine is a naturally occurring chemical involved in the production of energy in muscle. Abnormalities in creatine have been linked to the progression of degenerative neuromuscular diseases such as amyotrophic lateral sclerosis (ALS, or Lou Gehrig's Disease). This study will test whether taking creatine can improve the symptoms of ALS.

DETAILED DESCRIPTION:
Amyotrophic lateral sclerosis is a progressive neurodegenerative disorder selectively affecting motor neurons, resulting in progressive weakness. Currently there is no known cure and a specific cause has not been identified. Creatine is a nutritional supplement that improves mitochondrial function and has been shown to protect motor neurons in animal models of ALS. Preliminary research indicates that creatine may also improve strength in patients with ALS. This study will determine the effect of creatine treatment on short-term muscle strength and long-term muscle deterioration in patients with ALS.

Participants in this study will be randomly assigned to receive either creatine or placebo. Participants will be enrolled in the study for 9 months. Quantitative muscle testing will be done weekly for the first 3 weeks; participants will then be followed monthly for the next 4 months and bimonthly for the remainder of the 9-month study. The study will also monitor purposeful exercise to determine if this enhances the benefit of creatine usage on muscle strength. Pulmonary function testing will accompany the muscle testing to determine if creatine strengthens respiratory muscles, thereby enhancing pulmonary function.

ELIGIBILITY:
Inclusion Criteria

* Diagnosis of probable or definite ALS
* At least 5 of 10 testable upper extremity muscle groups (shoulder and elbow extensors/flexors and grip) of Medical Research Council (MRC) grade 4 or better
* At least 5 years from onset of symptoms

Exclusion Criteria

* Requires tracheostomy ventilation
* History of renal disease

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110
Dates: Start 2002-12; Study Completion 2006-05

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Rosenfeld, MD, Principal Investigator — Carolinas Medical Center
Locations (6):
- United States (6):
  - California Pacific Medical Center, San Francisco, California
  - Rush-Presbyterian St. Luke's Medical Center, Chicago, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - University of New Mexico - Medical Center, Albuquerque, New Mexico
  - University of Texas Health and Science Center, San Antonio, Texas
  - University of Virginia Health System, Charlottesville, Virginia